CLINICAL TRIAL: NCT00591266
Title: A Double-Blind, Randomized, Placebo-Controlled Study to Evaluate the Efficacy and Safety of TAK-491 When Co-administered With Amlodipine 5 mg in Subjects With Essential Hypertension
Brief Title: Efficacy and Safety of Azilsartan Medoxomil, Once Daily (QD), Co-Administered With Amlodipine in Participants With Essential Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sr. VP, Clinical Science, Takeda Global Research & Development Center, Inc.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 01-05-TL-491-010; U1111-1113-9132 (Registry Identifier: WHO)
Record Dates: First submitted 2007-12-27; First posted 2008-01-11 (Estimated); Results first posted 2011-04-19 (Estimated); Last update posted 2011-07-22 (Estimated); Status verified 2011-07

CONDITIONS: Hypertension
Keywords: Blood pressure; blood pressure monitoring ambulatory; Drug Therapy
MeSH Terms: conditions — Hypertension | interventions — azilsartan medoxomil; Amlodipine; azilsartan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Azilsartan Medoxomil 40 mg QD and Amlodipine 5 mg QD (Experimental)
  Interventions: Drug: Azilsartan Medoxomil and amlodipine
- Azilsartan Medoxomil 80 mg QD and Amlodipine 5 mg QD (Experimental)
  Interventions: Drug: Azilsartan Medoxomil and amlodipine
- Amlodipine 5 mg QD (Active Comparator)
  Interventions: Drug: Amlodipine

INTERVENTIONS:
Drug: Azilsartan Medoxomil and amlodipine — Azilsartan Medoxomil 40 mg, tablets, orally, once daily and amlodipine 5 mg, tablets, orally, once daily for up to 6 weeks.
  Other Names: Norvasc; TAK-491; Edarbi
  Arms: Azilsartan Medoxomil 40 mg QD and Amlodipine 5 mg QD
Drug: Azilsartan Medoxomil and amlodipine — Azilsartan Medoxomil 80 mg, tablets, orally, once daily and amlodipine 5 mg, tablets, orally, once daily for up to 6 weeks.
  Other Names: Norvasc; TAK-491; Edarbi
  Arms: Azilsartan Medoxomil 80 mg QD and Amlodipine 5 mg QD
Drug: Amlodipine — Azilsartan medoxomil placebo-matching tablets, orally, once daily and amlodipine 5 mg, tablets, orally, once daily for up to 6 weeks.
  Other Names: Norvasc
  Arms: Amlodipine 5 mg QD

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of azilsartan medoxomil, once daily (QD), co-administered with amlodipine in treating individuals with essential hypertension, compared to treatment with amlodipine alone.

DETAILED DESCRIPTION:
Hypertension affects approximately 50 million individuals in the United States. As the population ages, the prevalence of hypertension will continue to increase if broad and effective preventive measures are not implemented. According to the World Health Organization, hypertension is the most common attributable cause of preventable death in developed nations, as uncontrolled hypertension greatly increases the risk of cardiovascular disease, cerebrovascular disease, and renal failure. Despite the availability of antihypertensive treatments, hypertension remains inadequately controlled; only about one third of patients continue to maintain control successfully.

A major component of blood pressure regulation is the renin-angiotensin-aldosterone system, a system of hormone-mediated feedback interactions that results in the relaxation or constriction of blood vessels in response to various stimuli. Angiotensin II, a polypeptide hormone, is formed from angiotensin I in a reaction catalyzed by angiotensin-converting enzyme as part of the renin-angiotensin-aldosterone system. Angiotensin II is the principal pressor agent of the renin-angiotensin-aldosterone system with a myriad of effects on the cardiovascular system and on electrolyte homeostasis.

Takeda Global Research & Development Center, Inc. is developing TAK-491 (azilsartan medoxomil) to treat patients with essential hypertension. Azilsartan medoxomil is a prodrug that is hydrolyzed to the active moiety, azilsartan, which is a selective antagonist of the angiotensin II type 1 receptor subtype.

Amlodipine is a slow-channel blocker that inhibits the transmembrane influx of calcium ions into vascular smooth muscle and cardiac muscle. It is a peripheral arterial vasodilator that acts directly on vascular smooth muscle to cause a reduction in peripheral vascular resistance and reduction in blood pressure.

This study is being conducted to determine whether administration of azilsartan medoxomil in combination with amlodipine in participants with uncontrolled hypertension is more efficacious in reducing systolic blood pressure than amlodipine alone. Participation in this study is anticipated to be approximately 10 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Has essential hypertension and 24-hour mean systolic blood pressure greater than or equal to 140 mm Hg and less than or equal to 180 mm Hg.
2. Females of childbearing potential who are sexually active must agree to use adequate contraception, and can neither be pregnant nor lactating from Screening throughout the duration of the study
3. Has clinical laboratory evaluations within the reference range for the testing laboratory or the results are deemed not clinically significant for inclusion into this study by the investigator.
4. Is willing to discontinue current antihypertensive medications.

Exclusion Criteria:

1. Has sitting trough clinic diastolic blood pressure greater than 119 mm Hg.
2. Has a baseline 24 hour ambulatory blood pressure monitoring reading of insufficient quality.
3. The subject is hypersensitive to angiotensin II receptor blockers or calcium channel blockers.
4. Has a recent history of myocardial infarction, heart failure, unstable angina, coronary artery bypass graft, percutaneous coronary intervention, hypertensive encephalopathy, cerebrovascular accident, or transient ischemic attack.
5. Has clinically significant cardiac conduction defects.
6. Has hemodynamically significant left ventricular outflow obstruction due to aortic valvular disease.
7. Has secondary hypertension of any etiology
8. Is non-compliant with study medication during placebo run-in period.
9. Has severe renal dysfunction or disease.
10. Has known or suspected unilateral or bilateral renal artery stenosis.
11. Has a history of drug abuse or a history of alcohol abuse within the past 2 years.
12. Has a previous history of cancer that has not been in remission for at least 5 years prior to the first dose of study drug.
13. Has type 1 or poorly controlled type 2 diabetes mellitus.
14. Has hyperkalemia as defined by the central laboratory normal reference range,
15. Has an alanine aminotransferase level of greater than 2.5 times the upper limit of normal, active liver disease or jaundice.
16. Has an upper arm circumference less than 24 cm or greater than 42 cm.
17. Works night (3rd) shift.
18. Currently participating in another investigational study or has participated in an investigational study within 30 days prior to randomization.
19. Has any other serious disease or condition that would compromise subject safety or make it difficult to successfully manage and follow the subject according to the protocol.
20. Has been randomized in a previous TAK-491 study.
21. Is required to take or continues taking any disallowed medication, prescription medication, herbal treatment or over-the counter medication that may interfere with evaluation of the study medication.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 566 (Actual)
Dates: Start 2007-10; Primary Completion 2009-03 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Executive Medical Director Clinical Science, Study Director — Takeda
Locations (50):
- United States (50):
  - Mesa, Arizona
  - Phoenix, Arizona
  - Anaheim, California
  - Beverly Hills, California
  - Burbank, California
  - Burlingame, California
  - La Jolla, California
  - Orange, California
  - Roseville, California
  - Tustin, California
  - Wheat Ridge, Colorado
  - Newark, Delaware
  - Washington D.C., District of Columbia
  - Hialeah, Florida
  - Longwood, Florida
  - Tampa, Florida
  - Honolulu, Hawaii
  - Boise, Idaho
  - Chicago, Illinois
  - Gurnee, Illinois
  - Peoria, Illinois
  - Elkhart, Indiana
  - Crestview Hills, Kentucky
  - Lexington, Kentucky
  - Riverdale, Maryland
  - Brockton, Massachusetts
  - Haverhill, Massachusetts
  - North Dartmouth, Massachusetts
  - Kansas City, Missouri
  - Omaha, Nebraska
  - Raleigh, North Carolina
  - Akron, Ohio
  - Canton, Ohio
  - Cincinnati, Ohio
  - Mogadore, Ohio
  - Norman, Oklahoma
  - Tulsa, Oklahoma
  - Warminster, Pennsylvania
  - Cumberland, Rhode Island
  - Arlington, Texas
  - Austin, Texas
  - Carrollton, Texas
  - Dallas, Texas
  - Houston, Texas
  - Irvine, Texas
  - Lake Jackson, Texas
  - North Richland Hills, Texas
  - Manassas, Virginia
  - Renton, Washington
  - Menomonee Falls, Wisconsin

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants enrolled at 65 investigative sites in Argentina, Chile, Mexico, Peru and the United States from 03 October 2007 to 03 April 2009.
Pre-assignment Details: Participants with uncontrolled hypertension were enrolled in one of three, once-daily (QD) treatment groups.
Groups:
- Azilsartan Medoxomil 40 mg QD Amlodipine 5 mg QD: Azilsartan Medoxomil 40 mg, tablets, orally, once daily and amlodipine 5 mg, tablets, orally, once daily for up to 6 weeks.
- Azilsartan Medoxomil 80 mg QD and Amlodipine 5 mg QD: Azilsartan Medoxomil 80 mg, tablets, orally, once daily and amlodipine 5 mg, tablets, orally, once daily for up to 6 weeks.
- Amlodipine 5 mg QD: Amlodipine 5 mg, tablets, orally, once daily for up to 6 weeks.
Period: Overall Study
Arm/Group | Azilsartan Medoxomil 40 mg QD Amlodipine 5 mg QD | Azilsartan Medoxomil 80 mg QD and Amlodipine 5 mg QD | Amlodipine 5 mg QD
Started | 189 (Randomized only) | 188 (Randomized only) | 189 (Randomized only)
Completed | 180 | 177 | 175
Not Completed | 9 | 11 | 14
Not completed — Adverse Event | 2 | 2 | 3
Not completed — Lost to Follow-up | 0 | 1 | 0
Not completed — Protocol Violation | 0 | 0 | 1
Not completed — Withdrawal by Subject | 6 | 2 | 5
Not completed — Lack of Efficacy | 0 | 2 | 0
Not completed — Other | 1 | 4 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Azilsartan Medoxomil 40 mg QD Amlodipine 5 mg QD | Azilsartan Medoxomil 80 mg QD and Amlodipine 5 mg QD | Amlodipine 5 mg QD | Total
Number analyzed (Participants) | 189 | 188 | 189 | 566
Age Categorical [Number; unit: participants]
  <45 years | 28 | 23 | 15 | 66
  Between 45 and 64 years | 97 | 111 | 115 | 323
  ≥65 years | 64 | 54 | 59 | 177
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 99 | 85 | 95 | 279
  Male | 90 | 103 | 94 | 287

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the 24-hour Mean Systolic Blood Pressure Measured by Ambulatory Blood Pressure Monitoring.
Description: The change in 24-hour mean systolic blood pressure measured at week 6 relative to baseline. Ambulatory blood pressure monitoring measures blood pressure at regular intervals throughout the day and night. The 24-hour mean is the average of all measurements recorded for 24 hours after dosing.
Time Frame: Baseline and Week 6.
Population: Full Analysis Set.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Azilsartan Medoxomil 40 mg QD Amlodipine 5 mg QD | Azilsartan Medoxomil 80 mg QD and Amlodipine 5 mg QD | Amlodipine 5 mg QD
Number analyzed (Participants) | 165 | 166 | 166
mmHg | -24.79 (0.757) | -24.51 (0.754) | -13.60 (0.754)
Statistical Analysis 1: Comparison: Azilsartan Medoxomil 40 mg QD Amlodipine 5 mg QD vs Amlodipine 5 mg QD; Test type: Superiority or Other; p < 0.001, ANCOVA — Postbaseline P-value was from ANCOVA with terms for treatment (as a factor) and baseline value (as a covariate). Unadjusted p-value is presented. Overall 0.05 level of significance for multiple comparisons controlled using closed testing procedure; Mean Difference (Final Values) = -11.19, 95% CI 2-sided [-13.29 to -9.09]
Statistical Analysis 2: Comparison: Azilsartan Medoxomil 80 mg QD and Amlodipine 5 mg QD vs Amlodipine 5 mg QD; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -10.91, 95% CI 2-sided [-13.00 to -8.81]

2. Secondary Outcome: Change From Baseline in Mean Trough Clinic Sitting Systolic Blood Pressure.
Description: The change in mean trough clinic sitting systolic blood pressure measured at final visit or week 6 relative to baseline. Systolic blood pressure is the arithmetic mean of the 3 trough sitting systolic blood pressure measurements.
Time Frame: Baseline and Week 6.
Population: Full analysis set with last observation carried forward.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Azilsartan Medoxomil 40 mg QD Amlodipine 5 mg QD | Azilsartan Medoxomil 80 mg QD and Amlodipine 5 mg QD | Amlodipine 5 mg QD
Number analyzed (Participants) | 187 | 183 | 179
mmHg | -26.96 (1.037) | -25.50 (1.048) | -15.94 (1.060)
Statistical Analysis 1: Comparison: Azilsartan Medoxomil 40 mg QD Amlodipine 5 mg QD vs Amlodipine 5 mg QD; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -11.02, 95% CI 2-sided [-13.93 to -8.10]
Statistical Analysis 2: Comparison: Azilsartan Medoxomil 80 mg QD and Amlodipine 5 mg QD vs Amlodipine 5 mg QD; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -9.56, 95% CI 2-sided [-12.48 to -6.63]

3. Secondary Outcome: Change From Baseline in the 24-hour Mean Diastolic Blood Pressure Measured by Ambulatory Blood Pressure Monitoring.
Description: The change in 24-hour mean diastolic blood pressure measured at week 6 relative to baseline. Ambulatory blood pressure monitoring measures blood pressure at regular intervals throughout the day and night. The 24-hour mean is the average of all measurements recorded for 24 hours after dosing.
Time Frame: Baseline and Week 6.
Population: Full Analysis Set.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Azilsartan Medoxomil 40 mg QD Amlodipine 5 mg QD | Azilsartan Medoxomil 80 mg QD and Amlodipine 5 mg QD | Amlodipine 5 mg QD
Number analyzed (Participants) | 165 | 166 | 166
mmHg | -15.26 (0.492) | -15.43 (0.490) | -7.79 (0.490)
Statistical Analysis 1: Comparison: Azilsartan Medoxomil 40 mg QD Amlodipine 5 mg QD vs Amlodipine 5 mg QD; Test type: Superiority or Other; p < 0.001, ANCOVA — Postbaseline P-value was from ANCOVA with terms for treatment (as a factor) and baseline value (as a covariate). Unadjusted p-value is presented; Mean Difference (Final Values) = -7.48, 95% CI 2-sided [-8.84 to -6.11]
Statistical Analysis 2: Comparison: Azilsartan Medoxomil 80 mg QD and Amlodipine 5 mg QD vs Amlodipine 5 mg QD; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -7.65, 95% CI 2-sided [-9.01 to -6.28]

4. Secondary Outcome: Change From Baseline in Mean Trough Clinic Sitting Diastolic Blood Pressure
Description: The change in mean trough clinic sitting diastolic blood pressure measured at final visit or week 6 relative to baseline. Diastolic blood pressure is the arithmetic mean of the 3 trough sitting diastolic blood pressure measurements.
Time Frame: Baseline and Week 6.
Population: Full analysis set with last observation carried forward.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Azilsartan Medoxomil 40 mg QD Amlodipine 5 mg QD | Azilsartan Medoxomil 80 mg QD and Amlodipine 5 mg QD | Amlodipine 5 mg QD
Number analyzed (Participants) | 187 | 183 | 179
mmHg | -12.00 (0.602) | -12.65 (0.609) | -7.07 (0.616)
Statistical Analysis 1: Comparison: Azilsartan Medoxomil 40 mg QD Amlodipine 5 mg QD vs Amlodipine 5 mg QD; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -4.93, 95% CI 2-sided [-6.62 to -3.23]
Statistical Analysis 2: Comparison: Azilsartan Medoxomil 80 mg QD and Amlodipine 5 mg QD vs Amlodipine 5 mg QD; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -5.58, 95% CI 2-sided [-7.28 to -3.88]

5. Secondary Outcome: Change From Baseline in Daytime (6am to 10 pm) Mean Systolic Blood Pressure Measured by Ambulatory Blood Pressure Monitoring.
Description: The change in daytime (6am to 10pm) mean systolic blood pressure measured at week 6 relative to baseline. Ambulatory blood pressure monitoring measures blood pressure at regular intervals throughout the day and night. Daytime mean is the average of all measurements recorded between the hours of 6 am and 10 pm.
Time Frame: Baseline and Week 6.
Population: Full Analysis Set.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Azilsartan Medoxomil 40 mg QD Amlodipine 5 mg QD | Azilsartan Medoxomil 80 mg QD and Amlodipine 5 mg QD | Amlodipine 5 mg QD
Number analyzed (Participants) | 165 | 166 | 166
mmHg | -25.42 (0.802) | -24.95 (0.800) | -13.79 (0.799)
Statistical Analysis 1: Comparison: Azilsartan Medoxomil 40 mg QD Amlodipine 5 mg QD vs Amlodipine 5 mg QD; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -11.64, 95% CI 2-sided [-13.86 to -9.41]
Statistical Analysis 2: Comparison: Azilsartan Medoxomil 80 mg QD and Amlodipine 5 mg QD vs Amlodipine 5 mg QD; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -11.17, 95% CI 2-sided [-13.39 to -8.95]

6. Secondary Outcome: Change From Baseline in Daytime (6am to 10 pm) Mean Diastolic Blood Pressure Measured by Ambulatory Blood Pressure Monitoring.
Description: The change in daytime (6am to 10pm) mean diastolic blood pressure measured at week 6 relative to baseline. Ambulatory blood pressure monitoring measures blood pressure at regular intervals throughout the day and night. Daytime mean is the average of all measurements recorded between the hours of 6 am and 10 pm.
Time Frame: Baseline and Week 6.
Population: Full Analysis Set.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Azilsartan Medoxomil 40 mg QD Amlodipine 5 mg QD | Azilsartan Medoxomil 80 mg QD and Amlodipine 5 mg QD | Amlodipine 5 mg QD
Number analyzed (Participants) | 165 | 166 | 166
mmHg | -15.81 (0.535) | -15.86 (0.533) | -7.82 (0.533)
Statistical Analysis 1: Comparison: Azilsartan Medoxomil 40 mg QD Amlodipine 5 mg QD vs Amlodipine 5 mg QD; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -7.99, 95% CI 2-sided [-9.47 to -6.50]
Statistical Analysis 2: Comparison: Azilsartan Medoxomil 80 mg QD and Amlodipine 5 mg QD vs Amlodipine 5 mg QD; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -8.04, 95% CI 2-sided [-9.52 to -6.55]

7. Secondary Outcome: Change From Baseline in the Nighttime (12 am to 6 am) Mean Systolic Blood Pressure Measured by Ambulatory Blood Pressure Monitoring.
Description: The change in nighttime (12am to 6am) mean systolic blood pressure measured at week 6 relative to baseline. Ambulatory blood pressure monitoring measures blood pressure at regular intervals throughout the day and night. Nighttime mean is the average of all measurements recorded between the hours of 12 am and 6 am.
Time Frame: Baseline and Week 6.
Population: Full Analysis Set.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Azilsartan Medoxomil 40 mg QD Amlodipine 5 mg QD | Azilsartan Medoxomil 80 mg QD and Amlodipine 5 mg QD | Amlodipine 5 mg QD
Number analyzed (Participants) | 165 | 166 | 166
mmHg | -22.75 (0.853) | -22.72 (0.849) | -13.05 (0.848)
Statistical Analysis 1: Comparison: Azilsartan Medoxomil 40 mg QD Amlodipine 5 mg QD vs Amlodipine 5 mg QD; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -9.70, 95% CI 2-sided [-12.07 to -7.34]
Statistical Analysis 2: Comparison: Azilsartan Medoxomil 80 mg QD and Amlodipine 5 mg QD vs Amlodipine 5 mg QD; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -9.67, 95% CI 2-sided [-12.03 to -7.31]

8. Secondary Outcome: Change From Baseline in the Nighttime (12 am to 6 am) Mean Diastolic Blood Pressure Measured by Ambulatory Blood Pressure Monitoring.
Description: The change in nighttime (12am to 6am) mean diastolic blood pressure measured at week 6 relative to baseline. Ambulatory blood pressure monitoring measures blood pressure at regular intervals throughout the day and night. Nighttime mean is the average of all measurements recorded between the hours of 12 am and 6 am.
Time Frame: Baseline and Week 6.
Population: Full Analysis Set.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Azilsartan Medoxomil 40 mg QD Amlodipine 5 mg QD | Azilsartan Medoxomil 80 mg QD and Amlodipine 5 mg QD | Amlodipine 5 mg QD
Number analyzed (Participants) | 165 | 166 | 166
mmHg | -13.76 (0.606) | -13.78 (0.604) | -7.50 (0.604)
Statistical Analysis 1: Comparison: Azilsartan Medoxomil 40 mg QD Amlodipine 5 mg QD vs Amlodipine 5 mg QD; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -6.26, 95% CI 2-sided [-7.94 to -4.57]
Statistical Analysis 2: Comparison: Azilsartan Medoxomil 80 mg QD and Amlodipine 5 mg QD vs Amlodipine 5 mg QD; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -6.28, 95% CI 2-sided [-7.96 to -4.60]

9. Secondary Outcome: Change From Baseline in the 12-hour Mean Systolic Blood Pressure Measured by Ambulatory Blood Pressure Monitoring
Description: The change in the 12-hour mean systolic blood pressure measured at week 6 relative to baseline. Ambulatory blood pressure monitoring measures blood pressure at regular intervals throughout the day and night. The 12-hour mean is the average of all measurements recorded in the first 12 hours after dosing.
Time Frame: Baseline and Week 6.
Population: Full Analysis Set.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Azilsartan Medoxomil 40 mg QD Amlodipine 5 mg QD | Azilsartan Medoxomil 80 mg QD and Amlodipine 5 mg QD | Amlodipine 5 mg QD
Number analyzed (Participants) | 165 | 166 | 166
mmHg | -26.10 (0.850) | -25.40 (0.847) | -13.82 (0.846)
Statistical Analysis 1: Comparison: Azilsartan Medoxomil 40 mg QD Amlodipine 5 mg QD vs Amlodipine 5 mg QD; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -12.27, 95% CI 2-sided [-14.63 to -9.92]
Statistical Analysis 2: Comparison: Azilsartan Medoxomil 80 mg QD and Amlodipine 5 mg QD vs Amlodipine 5 mg QD; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -11.58, 95% CI 2-sided [-13.93 to -9.23]

10. Secondary Outcome: Change From Baseline in the 12-hour Mean Diastolic Blood Pressure Measured by Ambulatory Blood Pressure Monitoring
Description: The change in the 12-hour mean diastolic blood pressure measured at week 8 relative to baseline. Ambulatory blood pressure monitoring measures blood pressure at regular intervals throughout the day and night. The 12-hour mean is the average of all measurements recorded in the first 12 hours after dosing.
Time Frame: Baseline and Week 6.
Population: Full Analysis Set.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Azilsartan Medoxomil 40 mg QD Amlodipine 5 mg QD | Azilsartan Medoxomil 80 mg QD and Amlodipine 5 mg QD | Amlodipine 5 mg QD
Number analyzed (Participants) | 165 | 166 | 166
mmHg | -16.13 (0.575) | -15.97 (0.574) | -7.74 (0.574)
Statistical Analysis 1: Comparison: Azilsartan Medoxomil 40 mg QD Amlodipine 5 mg QD vs Amlodipine 5 mg QD; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -8.39, 95% CI 2-sided [-9.98 to -6.79]
Statistical Analysis 2: Comparison: Azilsartan Medoxomil 80 mg QD and Amlodipine 5 mg QD vs Amlodipine 5 mg QD; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -8.23, 95% CI 2-sided [-9.82 to -6.64]

11. Secondary Outcome: Change From Baseline in the Trough (22-24-hr) Mean Systolic Blood Pressure Measured by Ambulatory Blood Pressure Monitoring.
Description: The change in trough mean systolic blood pressure measured at week 6 relative to baseline. Ambulatory blood pressure monitoring measures blood pressure at regular intervals throughout the day and night. The trough mean is the average of all measurements recorded from 22 to 24 hours after dosing.
Time Frame: Baseline and Week 6.
Population: Full Analysis Set.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Azilsartan Medoxomil 40 mg QD Amlodipine 5 mg QD | Azilsartan Medoxomil 80 mg QD and Amlodipine 5 mg QD | Amlodipine 5 mg QD
Number analyzed (Participants) | 165 | 166 | 166
mmHg | -22.60 (0.942) | -22.67 (0.938) | -13.76 (0.938)
Statistical Analysis 1: Comparison: Azilsartan Medoxomil 40 mg QD Amlodipine 5 mg QD vs Amlodipine 5 mg QD; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -8.83, 95% CI 2-sided [-11.45 to -6.22]
Statistical Analysis 2: Comparison: Azilsartan Medoxomil 80 mg QD and Amlodipine 5 mg QD vs Amlodipine 5 mg QD; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -8.91, 95% CI 2-sided [-11.51 to -6.30]

12. Secondary Outcome: Change From Baseline in the Trough (22-24-hr) Mean Diastolic Blood Pressure Measured by Ambulatory Blood Pressure Monitoring.
Description: as for outcome 11
Time Frame: Baseline and Week 6.
Population: Full Analysis Set.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Azilsartan Medoxomil 40 mg QD Amlodipine 5 mg QD | Azilsartan Medoxomil 80 mg QD and Amlodipine 5 mg QD | Amlodipine 5 mg QD
Number analyzed (Participants) | 165 | 166 | 166
mmHg | -14.34 (0.698) | -14.93 (0.696) | -8.39 (0.696)
Statistical Analysis 1: Comparison: Azilsartan Medoxomil 40 mg QD Amlodipine 5 mg QD vs Amlodipine 5 mg QD; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -5.94, 95% CI 2-sided [-7.88 to -4.00]
Statistical Analysis 2: Comparison: Azilsartan Medoxomil 80 mg QD and Amlodipine 5 mg QD vs Amlodipine 5 mg QD; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -6.54, 95% CI 2-sided [-8.47 to -4.61]

13. Secondary Outcome: Percentage of Participants Who Achieve a Clinic Systolic Blood Pressure Response, Defined as < 140 mm Hg and/or Reduction From Baseline ≥ 20 mm Hg
Description: Percentage of participants who achieve a clinic systolic blood pressure response measured at week 6 relative to baseline, defined as less than 140 mm Hg and/or reduction from baseline of greater than or equal to 20 mm Hg. Systolic blood pressure is the arithmetic mean of the 3 trough sitting systolic blood pressure measurements.
Time Frame: Baseline and Week 6.
Population: Full analysis set with last observation carried forward.
Measure: Number; unit: percentage of participants
Arm/Group | Azilsartan Medoxomil 40 mg QD Amlodipine 5 mg QD | Azilsartan Medoxomil 80 mg QD and Amlodipine 5 mg QD | Amlodipine 5 mg QD
Number analyzed (Participants) | 187 | 183 | 179
percentage of participants | 72.7 | 71.6 | 45.8
Statistical Analysis 1: Comparison: Azilsartan Medoxomil 40 mg QD Amlodipine 5 mg QD vs Amlodipine 5 mg QD; Test type: Superiority or Other; p < 0.001, Regression, Logistic — P-value for response criteria for systolic blood pressure was from a logistic regression with treatment as a factor and baseline clinic systolic blood pressure as a covariate. The unadjusted p-value is presented; Odds Ratio (OR) = 3.37, 95% CI 2-sided [2.15 to 5.26]
Statistical Analysis 2: Comparison: Azilsartan Medoxomil 80 mg QD and Amlodipine 5 mg QD vs Amlodipine 5 mg QD; Test type: Superiority or Other; p < 0.001, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.21, 95% CI 2-sided [2.05 to 5.03]

14. Secondary Outcome: Percentage of Participants Who Achieve a Clinic Diastolic Blood Pressure Response, Defined as < 90 mm Hg and/or Reduction From Baseline ≥ 10 mm Hg
Description: Percentage of participants who achieve a clinic diastolic blood pressure response measured at week 6 relative to baseline, defined as less than 90 mm Hg and/or reduction from baseline of greater than or equal to 10 mm Hg. Diastolic blood pressure is the arithmetic mean of 3 trough sitting diastolic blood pressure measurements.
Time Frame: Baseline and Week 6.
Population: Full analysis set with last observation carried forward.
Measure: Number; unit: percentage of participants
Arm/Group | Azilsartan Medoxomil 40 mg QD Amlodipine 5 mg QD | Azilsartan Medoxomil 80 mg QD and Amlodipine 5 mg QD | Amlodipine 5 mg QD
Number analyzed (Participants) | 187 | 183 | 179
percentage of participants | 86.1 | 87.4 | 65.9
Statistical Analysis 1: Comparison: Azilsartan Medoxomil 40 mg QD Amlodipine 5 mg QD vs Amlodipine 5 mg QD; Test type: Superiority or Other; p < 0.001, Regression, Logistic — P-value for response criteria for diastolic blood pressure was from a logistic regression with treatment as a factor and baseline clinic diastolic blood pressure as a covariate. The unadjusted p-value is presented; Odds Ratio (OR) = 3.54, 95% CI 2-sided [2.08 to 6.02]
Statistical Analysis 2: Comparison: Azilsartan Medoxomil 80 mg QD and Amlodipine 5 mg QD vs Amlodipine 5 mg QD; Test type: Superiority or Other; p < 0.001, Regression, Logistic — [p-value comment as in outcome 14, analysis 1]; Odds Ratio (OR) = 3.90, 95% CI 2-sided [2.25 to 6.75]

15. Secondary Outcome: Percentage of Participants Who Achieve Both a Clinic Diastolic and Systolic Blood Pressure Response
Description: Percentage of participants who achieve both a clinic diastolic and systolic blood pressure response measured at week 6 relative to baseline, defined as less than 90 mm Hg and/or reduction from baseline of greater than or equal to 10 mm Hg AND less than 140 mm Hg and/or reduction from baseline of greater than or equal to 20 mm Hg. Diastolic and systolic blood pressure is based on the arithmetic mean of the 3 sitting blood pressure measurements.
Time Frame: Baseline and Week 6.
Population: Full analysis set with last observation carried forward.
Measure: Number; unit: percentage of participants
Arm/Group | Azilsartan Medoxomil 40 mg QD Amlodipine 5 mg QD | Azilsartan Medoxomil 80 mg QD and Amlodipine 5 mg QD | Amlodipine 5 mg QD
Number analyzed (Participants) | 187 | 183 | 179
percentage of participants | 65.8 | 69.4 | 43.0
Statistical Analysis 1: Comparison: Azilsartan Medoxomil 40 mg QD Amlodipine 5 mg QD vs Amlodipine 5 mg QD; Test type: Superiority or Other; p < 0.001, Regression, Logistic — P-value for joint response criteria for systolic blood pressure and diastolic blood pressure was from a logistic regression with treatment as a factor and baseline clinic systolic blood pressure as a covariate. The unadjusted p-value is presented; Odds Ratio (OR) = 2.62, 95% CI 2-sided [1.71 to 4.02]
Statistical Analysis 2: Comparison: Azilsartan Medoxomil 80 mg QD and Amlodipine 5 mg QD vs Amlodipine 5 mg QD; Test type: Superiority or Other; p < 0.001, Regression, Logistic — [p-value comment as in outcome 15, analysis 1]; Odds Ratio (OR) = 3.12, 95% CI 2-sided [2.01 to 4.82]

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events are adverse events that started after the first dose of double-blind study drug and no more than 14 days (or 30 days for a serious adverse event) after the last dose of double-blind study drug.
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Azilsartan Medoxomil 40 mg QD Amlodipine 5 mg QD | Azilsartan Medoxomil 80 mg QD and Amlodipine 5 mg QD | Amlodipine 5 mg QD
Serious Adverse Events (participants affected / at risk) | 1/190 | 2/188 | 1/185
Other Adverse Events (participants affected / at risk) | 11/190 | 10/188 | 10/185
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Azilsartan Medoxomil 40 mg QD Amlodipine 5 mg QD (N=190) | Azilsartan Medoxomil 80 mg QD and Amlodipine 5 mg QD (N=188) | Amlodipine 5 mg QD (N=185)
Chest pain (General disorders) | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0
Ovarian cyst torsion (Reproductive system and breast disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Azilsartan Medoxomil 40 mg QD Amlodipine 5 mg QD (N=190) | Azilsartan Medoxomil 80 mg QD and Amlodipine 5 mg QD (N=188) | Amlodipine 5 mg QD (N=185)
Headache (Nervous system disorders) | 11 | 10 | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No publication related to study results will be published prior to publication of a multi-center report submitted for publication within 18 months after conclusion or termination of a study at all study sites. Results publications will be submitted to sponsor for review 60 days in advance of publication. Sponsor can require removal of confidential information unrelated to study results. Sponsor can embargo a proposed publication for another 60 days to preserve intellectual property.